CLINICAL TRIAL: NCT03353844
Title: The Effects of Intradialytic Exercise on Daily Physical Activity in Patients Undergoing Long-term High-efficiency Online Hemodiafiltration
Brief Title: The Effects of Intradialytic Exercise in Hemodiafiltration Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khajohn Tiranathanagul, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 139/60
Record Dates: First submitted 2017-11-08; First posted 2017-11-27 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: End Stage Renal Disease; Hemodialysis; Sedentary Lifestyle
MeSH Terms: conditions — Kidney Failure, Chronic; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradialytic exercise group (Experimental): These patients will get intradialytic exercise every sessions of hemodiafiltration
  Interventions: Behavioral: Intradialytic exercise
- Standard dialysis group (No Intervention): regular and standard of care in every hemodiafiltration sessions (as usual) without intradialytic exercise.

INTERVENTIONS:
Behavioral: Intradialytic exercise — intradialytic exercise which start and finish in first hour of hemodiafiltration session
  Arms: Intradialytic exercise group

SUMMARY:
Low physical activity is associated with in hemodialysis and hemodiafiltration (HDF) patients. Previous studies showed the benefits of intradialytic exercise for improvement of physical fitness and hemodialysis adequacy. However, the effect of intradialytic exercise on physical activity has not been explored. This current open-labelled randomized controlled trial is conducted in HDF patients to determine the effect of intradialytic exercise program for 6 months on daily physical activity measured by tri-axial accelerometer (wearable device).

DETAILED DESCRIPTION:
The study is an open-labelled randomized controlled trial which compare the changes of daily physical activity measured by tri-axial accelerometer (wearable device) between the HDF patients in intradialytic exercise group and control during the 6-month period. After inclusion in to the study, all of the participants will be evaluated before randomized. The investigators will prescribe the exercise program for each participant in the exercise group. The exercise program use intradialytic cycling which will be gradually increased to at least 30 minutes with moderate intensity. The participants in control group will receive dialysis as usual without intradialytic exercise prescription. The participants will go on the program for at least 6-months period. In each session, any adverse event or side effect will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis vintage more than 3 months
* Sedentary or light physical activity

Exclusion Criteria:

* recent myocardial infarction (<12 months)
* recent ischemic stroke (<12months)
* uncontrolled comorbidities (diabetes/hypertension/heart failure/heart disease/respiratory disease)
* Life expectancy < 12 months
* active musculoskeletal problem e.g.) rheumatoid arthritis, spondyloarthropathy, osteoarthritis, fracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Change of daily physical activity at 6 months | at 0 and 6 months
  Every participant will be monitored their daily physical activity by wearable tri-axial accelerometer (Fitbit) before and at 6 months to observe changes in daily physical activity.

SECONDARY OUTCOMES:
Dialysis adequacy as measured by kt/V | at 6 months
  Adequacy of dialysis will be monitor at baseline and 6 month
Aerobic exercise capacity as measured by VO2 max | at 6 months
  Aerobic exercise capacity parameters including VO2 max (maximal oxygen consumption) will be measured at baseline and 6 month
Body composition (lean and fat body mass) | at 6 months
  The baseline body composition measurements and body composition at 6 months will be measured by DXA scan and bioimpedance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Khajohn Tiranathanagul, MD, Principal Investigator — Chulalongkorn University; Nawaporn Assawasaksakul, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Derived] Assawasaksakul N, Sirichana W, Joosri W, Kulaputana O, Eksakulkla S, Ketanun C, Kittiskulnam P, Chantadisai M, Takkavatakarn K, Susantitaphong P, Praditpornsilpa K, Eiam-Ong S, Tiranathanagul K. Effects of intradialytic cycling exercise on daily physical activity, physical fitness, body composition, and clinical parameters in high-volume online hemodiafiltration patients: a pilot randomized-controlled trial. Int Urol Nephrol. 2021 Feb;53(2):359-371. doi: 10.1007/s11255-020-02677-7. Epub 2020 Oct 31. PMID 33128722